CLINICAL TRIAL: NCT05385341
Title: Is Tele-rehabilitation an Efficacious Alternative to Traditional Center Based Cardiac Rehabilitation After Acute Coronary Syndrome?
Brief Title: Rehabilitation Exercise with MObile Technology and Education After Acute Coronary Syndrome
Acronym: REMOTE-ACS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The start of the study took too long and there are already many publications on the subject
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/18/0474
Record Dates: First submitted 2020-04-21; First posted 2022-05-23 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Acute Coronary Syndrome
Keywords: Cardiac rehabilitation; Tele-health
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Telerehabilitation; Rehabilitation; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation (Tele RCV) (Experimental): Experimental group (Tele-RCV): the treatment will consist of 20 home-based sessions monitored by the REMOTE-ACS device and containing 2 hours/day 5 days/7 of exercise training (the first session in center to form the patient) associated with 8 educative sessions.
  Interventions: Other: Telerehabilitation (Tele RCV)
- Rehabilitation (RCV) (Active Comparator): Group control (RCV) : 20 sessions of cardiac rehabilitation will be realized in a rehabilitation center containing exercise training during 2 hours/day 5 days/7 and educative program.
  Interventions: Other: Rehabilitation (RCV)

INTERVENTIONS:
Other: Telerehabilitation (Tele RCV) — 20 home-based sessions monitored by the REMOTE-ACS device and containing 2 hours/day 5 days/7 of exercise training associated with educative sessions.
  Arms: Telerehabilitation (Tele RCV)
Other: Rehabilitation (RCV) — 20 sessions of cardiac rehabilitation will be realized in a rehabilitation center containing exercise training during 2 hours/day 5 days/7 and educative program.
  Arms: Rehabilitation (RCV)

SUMMARY:
Despite a clear indication of grade Ia, cardiac rehabilitation (CR) is dramatically underutilized after acute coronary syndrome with less than 30% of patients addressed in France. Mobile technology has the potential to overcome barriers to access to cardiac rehabilitation and may be a useful tool for increasing participation. However, studies have to prove this type of care is as effective as traditional center based cardiac rehabilitation.

DETAILED DESCRIPTION:
After acute coronary syndrome (ACS), it is recommended to propose a cardiac rehabilitation (CR) program in order to reduce the risk of recidive, to improve the quality of life and to reduce the risk of disabilities. Traditional CR which is most of the time center-based, is underutilized with less than 30% of patients addressed en France. Therefore, Télé-Cardiac Rehabilitation (Télé-RCV) has been developped progressively since the eighties showing comparable efficacity compared with CR concerning physical fitness. The investigative team, had previously published results showing that telephone support guided by accelerometers could improve physical activity. However, In France, device allowing telemonitoring online of heart rate are not available. Moreover, the investigators have not yet developped remote therapeutic education which is proposed in CR programs. Thus, the present study planned to develop and evaluate aTele-RCV solution aimed to monitor exercise training at home and to educate remotely patient after ACS.

The device is an association of a heart rate monitor, a blood pressure testing, a balance linked with a full web secured application connecting patient and caregivers. In the intervention group, Tele-RCV is proposed during 20 sessions containing 2h of exercise training combined with 6h of therapeutic tele-education. In the control group, CR is proposed during 20 sessions with the same volume of exercise training and therapeutic education. After randomisation, patient are allocated to one of the two groups. The evaluation of the primary and secondary outcomes are realized at the beginning, at one month (only walking tests) and at 2 months. A social evaluation is done in parallel to test the acceptability for the Télé-RCV compared with CR.

ELIGIBILITY:
Inclusion Criteria:

* Patient with acute coronary syndrome less than 6 months,
* Addressed to ambulatory cardiac rehabilitation,
* Equipped with a smartphone compatible with the protocol's application, connected to web
* Having signed an informed consent,
* Affiliated to the french national health insurance.

Exclusion Criteria:

* Incapacity to use application on smartphone,
* Contraindication to exercise training,
* Pregnancy,
* Juridic protection
* Left ventricular ejection fraction < 45%
* Significate ventricular arrhythmia (frequent or polymorph PVC during initial exercise testing, ventricular tachycardia or sudden cardiac death at the beginning)
* Flutter or atrial fibrillation (transient or permanent)
* Coronary revascularization needing supplementary procedure
* Residual myocardial ischemia determined by initial exercise testing or alternative testing (nuclear imaging or stress echocardiography)
* Mini Mental State < 26
* Patients living alone at home
* Comorbidities limiting participation to the protocol: kidney dialysis, insulin-requiring diabetes, residuals sequels of central and/or peripheral nervous system injuries

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect analysis 2 month after inclusion | 2 months
  Change of the peak oxygen volume at 2 months after inclusion

SECONDARY OUTCOMES:
Effect analysis 1 month after inclusion | 1 month
  Analysis of change between T0 and 1 month concerning the walking tests : distance traveled in meters
Effect analysis 1 month after inclusion | 1 month
  Analysis of change between T0 and 1 month concerning the number of Tele-RCV or RCV sessions realized
Effect analysis 2 months after inclusion | 2 months
  Analysis of change between T0 and 2 months concerning the walking tests:distance traveled in meters
Effect analysis 2 months after inclusion | 2 months
  Analysis of change between T0 and 2 months concerning the number of Tele-RCV or RCV sessions realized
Health economics criteria | 26 months
  Incremental Cost-effectiveness ratios of the REMOTE-ACS device compared with the traditional cardiac rehabilitation after acute coronary syndrome according to the French national health insurance perspective and 2 months follow-up period.
Health economics criteria | 26 months
  Cost-utility ratios of the REMOTE-ACS device compared with the traditional cardiac rehabilitation after acute coronary syndrome according to the French national health insurance perspective and 2 months follow-up period.
Production cost of the REMOTE-ACS device | 26 months
  Production cost of the REMOTE-ACS device by micro costing, according the hospital perspective
Acceptability of the device | 26 months
  The acceptability will be assessed by a sociological point of view based on collective meeting (with patient and caregivers) and individual questionnaires for the two groups before randomization and after the program only for the Tele-RCV group.
Satisfaction of the device | 26 months
  The satisfaction will be assessed by a questionnaire of satisfaction titled: Cardiovascular rehabilitation program satisfaction questionnaire, with 8 questions, the minimum value is "nothing", and the maximum value is "very important"

CONTACTS AND LOCATIONS:
Overall Officials: Meyer ELBAZ, MD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No